CLINICAL TRIAL: NCT01622257
Title: Comparison of Cavitation Ultrasound, Metformin or the Combination of Both in Obese Women With Polycystic Ovary Syndrome
Brief Title: Cavitation Ultrasound in Treatment of Patients With PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Lecturer, Ain Shams University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ASU6-2011
Record Dates: First submitted 2012-06-18; First posted 2012-06-19 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: PCOS
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cavitation US (Experimental): Cavitation ultrasound was done using ultrasonic cavitation machine 2 times per week for 3 months
  Interventions: Device: Cavitation US
- Metformin (Experimental): Metformin oral tablets 500 mg were given three times daily
  Interventions: Drug: Metformin
- Cavitation US + metformin (Experimental): Combination of both Cavitation US + Metformin
  Interventions: Other: Cavitation US + Metformin

INTERVENTIONS:
Device: Cavitation US — The areas with localized fat are treated 2 times per week for 3 months using Aesthetic cavitation via ultrasonic cavitation machine (Cavi SMART, South Korea, supplied with one piece cavitation probe of 40 KHz, 3-6 watt(W)/cm^2 adjustable, 60W with 20cm^2 active surface).
  Other Names: Cavi SMART
  Arms: Cavitation US
Drug: Metformin — Metformin hydrochloride (Glucophage 500 mg/tablet, Bristol-Myers Squibb, New York, USA). Medication is initiated in a step-up fashion every 5 days, from one tablet per day to three. This dose is maintained as tolerated throughout the 3 months of the study.
  Other Names: Glucophage, Bristol-Myers Squibb, New York, USA
  Arms: Metformin
Other: Cavitation US + Metformin — Combination of both Cavitation US + Metformin. the treatment duration lasts 3 months
  Other Names: Glucophage + Cavi SMART
  Arms: Cavitation US + metformin

SUMMARY:
The aim of the current work was to compare the efficacy of cavitation ultrasound, metformin or combination of both in obese women with polycystic ovary syndrome (PCOS) regarding clinical pregnancy rate, ovulation rate, insulin resistance, serum testosterone level, lipid profile.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 5 to 10% of women of childbearing age and is the most common cause of anovulatory infertility. Common clinical manifestations include menstrual irregularities and signs of androgen excess such as hirsutism, acne, and alopecia. Metformin, a biguanide, is the most widely used drug for the treatment of type 2 diabetes worldwide. Its primary action is to inhibit hepatic glucose production, but it also increases the sensitivity of peripheral tissues to insulin. The increase in insulin sensitivity, which contributes to the efficacy of metformin in the treatment of diabetes, has also been shown in non diabetic women with the polycystic ovary syndrome.In women with PCOS, long-term treatment with metformin may increase ovulation, improve menstrual cyclicity, and reduce serum androgen levels; the use of metformin may also improve hirsutism. If published data on the effects of metformin in the prevention of diabetes can be extrapolated to women with the PCOS, then the drug may actually retard progression to glucose intolerance in affected women, as reported in a small, retrospective study. Ultrasonic vibrations spread in the form of a wave in medium such as a liquid or a solid. When the particles of an elastic medium are under ultrasonic vibration, they act continuously in only one direction. The lipolytic range of ultrasounds is 30-70 Kilohertz (KHz), and the best effects are obtained in a range between30-35 KHz. The depth of the treatment in the tissues is generally2-3 cm, to avoid muscles involvement. Biological effects of ultrasounds on adipocytes are: micro-mechanical, thermal, micro-streaming and cavitation. Cavitation ultrasound means that ultrasounds produce an alternation of decompression and compression waves in a fluid media which progressively increase the tension of the adipocyte until it implodes and frees the emulsified fat. The aim of the current work was to compare the efficacy of cavitation ultrasound, metformin or combination of both in obese women with polycystic ovary syndrome (PCOS) regarding clinical pregnancy rate, ovulation rate, insulin resistance, serum testosterone level, lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Obese infertile polycystic ovarian syndrome (PCOS) women

Exclusion Criteria:

* Women 40 years or older
* Women using fertility treatments, oral contraceptives or other confounding medications during the last 3 months
* Smokers or with history of general diseases like cardiovascular, liver, kidney or respiratory disease, diabetes, uncontrolled hypertension, or malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa I. Ibrahem, M.D., Study Director — Ain Shams University; Mohamed I. Ellaithy, MD, Study Chair — Lecturer Obstetics & Gynecology Ain shams university faculty of medicine; Ahmed K. Makled, MD, Principal Investigator — Assistant professor of Obstetrics & Gynecology Ain shams university faculty of medicine
Locations (1):
- Ain shams university, Cairo, Egypt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 252 women were assessed for eligibility 54 women were excluded
  * Not meeting inclusion criteria (n=38)
  * Declined to participate (n=9)
  * Other reasons (n=7)
Groups:
- Metformin: Metformin oral tablets 500 mg were given three times daily for 3 months
Period: Overall Study
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin
Started | 66 | 66 | 66
Completed | 66 | 66 | 66
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin | Total
Number analyzed (Participants) | 66 | 66 | 66 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.7 (4.5) | 26.1 (4.1) | 26.3 (5.2) | 26 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 66 | 198
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Egypt | 66 | 66 | 66 | 198
Duration of infertility [Mean (Standard Deviation); unit: Years] | 3.3 (1.5) | 3.4 (1.3) | 3.2 (1.3) | 3.3 (1.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 37.9 (4.9) | 36.7 (4.2) | 36.1 (5.2) | 36.9 (4.7)
Androgenic alopecia [Number; unit: Participants]
  Yes | 12 | 9 | 6 | 27
  No | 54 | 57 | 60 | 171
Acne [Number; unit: Participants]
  Yes | 18 | 23 | 26 | 67
  No | 48 | 43 | 40 | 131
Seborrheic dermatitis [Number; unit: Participants]
  Yes | 26 | 34 | 39 | 99
  No | 40 | 32 | 27 | 99
Menstrual pattern [Number; unit: Participants]
  Amenorrhea | 43 | 47 | 51 | 141
  Oligomenorrhea | 23 | 19 | 15 | 57
Systolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 122.4 (10.1) | 121.9 (12.4) | 121.8 (12.3) | 122 (11.6)
Diastolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 80.5 (8.2) | 81.6 (7.1) | 82.9 (7.8) | 81.7 (7.6)
Serum Follicle-stimulating Hormone (FSH) [Mean (Standard Deviation); unit: mIU/ml] | 6.1 (1.9) | 5.8 (2.2) | 6.6 (2.3) | 6.2 (2.1)
Luteinizing Hormone (LH) [Mean (Standard Deviation); unit: mIU/ml] | 10.9 (1.1) | 10.7 (1.1) | 11.1 (1.8) | 10.9 (1.3)
LH/FSH ratio [Mean (Standard Deviation); unit: Ratio] | 1.79 (0.7) | 1.85 (0.6) | 1.68 (0.6) | 1.77 (0.6)
Total testosterone [Mean (Standard Deviation); unit: ng/ml] | 0.84 (0.05) | 0.83 (0.04) | 0.83 (0.04) | 0.83 (0.04)
Free testosterone [Mean (Standard Deviation); unit: pg/ml] | 3.9 (2.07) | 3.8 (1.32) | 3.7 (1.72) | 3.8 (1.71)
Fasting insulin [Mean (Standard Deviation); unit: µIU/ml] | 12.9 (6.4) | 12.5 (5.3) | 11.8 (4.1) | 12.4 (5.1)
Fasting glucose [Mean (Standard Deviation); unit: mg/dl] | 83.1 (21.4) | 79.4 (22.7) | 77.8 (22.1) | 80.1 (22.3)
Fasting Glucose/Insulin Ratio (GIR) [Mean (Standard Deviation); unit: mg/mIU] | 6.44 (0.8) | 6.35 (0.7) | 6.59 (0.7) | 6.46 (0.7)
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: HOMA score] — Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)= Fasting insulin x Fasting glucose / 22.5
  HOMA score | 2.65 (1.01) | 2.45 (1.06) | 2.27 (0.99) | 2.46 (1.01)
Quantitative Insulin sensitivity Check Index (QUICKI) [Mean (Standard Deviation); unit: Index] — The quantitative insulin sensitivity check index (QUICKI) is derived using the inverse of the sum of the logarithms of the fasting insulin and fasting glucose:
  1 / [(log(fasting insulin µU/mL) + log(fasting glucose mg/dL)]
  µU/mL, microunits/milliliter; mg/dL, milligrams/deciliter.
  Index | 0.33 (0.03) | 0.33 (0.04) | 0.34 (0.04) | 0.33 (0.04)
Total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 282.3 (32) | 273.4 (29.2) | 276.8 (30.5) | 277.2 (30.7)
Low-density lipoprotein (LDL) [Mean (Standard Deviation); unit: mg/dl] | 129.7 (19.3) | 127.1 (20.4) | 122.6 (19.1) | 126.5 (19.6)
High-density lipoprotein (HDL) [Mean (Standard Deviation); unit: mg/dl] | 80.9 (11.2) | 77.8 (9.9) | 82.1 (10.8) | 80.4 (10.6)
Triglycerides (TGs) [Mean (Standard Deviation); unit: mg/dl] | 204.9 (28.1) | 199.6 (22.4) | 208.4 (26.8) | 204.3 (25.7)
Waist to Hip Ratio (WHR) [Mean (Standard Deviation); unit: Ratio] | 0.88 (0.7) | 0.89 (0.7) | 0.91 (0.8) | 0.89 (0.7)
Total body fat percent [Mean (Standard Deviation); unit: Percentage] | 43.2 (5.6) | 44.9 (6.2) | 45.6 (5.7) | 44.6 (5.8)
Body fat mass [Mean (Standard Deviation); unit: Kilograms (kg)] | 37.7 (10.4) | 39.8 (11.2) | 41.1 (10.1) | 39.5 (10.5)
Fat free mass [Mean (Standard Deviation); unit: Kilograms (kg)] | 50.8 (9.5) | 51.2 (9.1) | 51.2 (10.2) | 51.1 (9.6)
Abdominal fat mass [Mean (Standard Deviation); unit: Kilograms (kg)] | 6.8 (2.8) | 6.9 (3.2) | 7.1 (2.2) | 6.9 (2.6)
Emotion mean score [Mean (Standard Deviation); unit: PCOSQ Emotion Score] — The Emotions score consists of 8 items:
  * Depressed
  * Easily tired
  * Moody
  * Had low self-esteem
  * Fear of getting cancer
  * Worried
  * Being self-conscious
  * Late menstrual period
  For each item there are seven rating options, 1 represents the greatest possible impairment, while 7 represents the least impairment.
  A 2-week time frame was chosen for patients to describe their function. PCOSQ Emotions mean score = the average of the 8 items (Range=1-7) (PCOSQ, The Polycystic Ovary Syndrome Questionnaire)
  PCOSQ Emotion Score | 4.3 (1.4) | 4.9 (1.6) | 4.7 (1.7) | 4.6 (1.6)
Body hair mean score [Mean (Standard Deviation); unit: PCOSQ Body hair Score] — The Body Hair score consists of 5 items:
  * Visible hair on chin
  * Visible hair on upper lip
  * Visible hair on face
  * Embarrassment about excessive body hair
  * Visible body hair
  For each item there are seven rating options, 1 represents the greatest possible impairment, while 7 represents the least impairment.
  A 2-week time frame was chosen for patients to describe their function. PCOSQ Body hair mean score = the average of the 5 items (Range=1-7) (PCOSQ, The Polycystic Ovary Syndrome Questionnaire)
  PCOSQ Body hair Score | 3.4 (1.7) | 3.3 (1.9) | 3.7 (1.6) | 3.5 (1.7)
Weight mean score [Mean (Standard Deviation); unit: PCOSQ Weight Score] — The Weight score consists of 5 items:
  * Concerned about being overweight
  * Trouble dealing with your weight
  * Frustration in losing weight
  * Do not feel sexy because of weight
  * Difficulties staying at ideal weight
  For each item there are seven rating options, 1 represents the greatest possible impairment, while 7 represents the least impairment.
  A 2-week time frame was chosen for patients to describe their function. PCOSQ Weight mean score = the average of the 5 items (Range=1-7) (PCOSQ, The Polycystic Ovary Syndrome Questionnaire)
  PCOSQ Weight Score | 2.6 (1.4) | 2.4 (1.3) | 2.1 (1.5) | 2.4 (1.4)
Menstrual problems mean score [Mean (Standard Deviation); unit: PCOSQ Menstrual problems Score] — The Menstrual problems score consists of 4 items:
  * Headaches
  * Irregular menstrual periods
  * Abdominal Bloating
  * Menstrual cramps
  For each item there are seven rating options, 1 represents the greatest possible impairment, while 7 represents the least impairment.
  A 2-week time frame was chosen for patients to describe their function. PCOSQ Menstrual problems mean score = the average of the 4 items (Range=1-7) (PCOSQ, The Polycystic Ovary Syndrome Questionnaire)
  PCOSQ Menstrual problems Score | 3.6 (1.1) | 3.7 (1.1) | 3.9 (1.1) | 3.7 (1.1)
Infertility mean score [Mean (Standard Deviation); unit: PCOSQ Infertility Score] — The Infertility score consists of 4 items:
  * Concerned with infertility problems
  * Fear of not having children
  * Feel lack of control over the situation
  * Sadness because of infertility problems
  For each item there are seven rating options, 1 represents the greatest possible impairment, while 7 represents the least impairment.
  A 2-week time frame was chosen for patients to describe their function. PCOSQ Infertility mean score = the average of the 4 items (Range=1-7) (PCOSQ, The Polycystic Ovary Syndrome Questionnaire)
  PCOSQ Infertility Score | 3.7 (1.02) | 3.6 (0.9) | 3.4 (1.1) | 3.6 (1)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin
Number analyzed (Participants) | 66 | 66 | 66
participants | 12 | 5 | 16

2. Secondary Outcome: Ovulation Rate as Determined by Ultrasonographic Folliculometry and Luteal Serum Progesterone Assay.
Description: The Number of participants who had evidence of successful ovulation during the 3 months. Ovulation was diagnosed based on ultrasonographic folliculometry and/or luteal serum progesterone assay.Every month, folliculometry was done to count the number of antral follicles (AFC), follow follicular growth, measure dominant follicle diameter and detect occurrence of ovulation. a mid-luteal serum progesterone assay was done to confirm ovulation.
  Ultrasound was performed serially till reaching preovulatory follicle(s of around 20 mm in diameter that then rupture to show a collapsed follicle in the same location with internal echoes consistent with its transformation to a corpus luteum. Progesterone assay was done using immulite 2000 apparatus chemiluminescent immunometric assay. Mid-luteal phase progesterone above 6 ng/mL was considered indicative of normal corpus. luteum function.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin
Number analyzed (Participants) | 66 | 66 | 66
participants | 39 | 16 | 45

3. Secondary Outcome: Change in Insulin Resistance
Description: Change in Fasting insulin concentration
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: uIU/ml
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin
Number analyzed (Participants) | 66 | 66 | 66
uIU/ml | -2.4 [-2.61 to -2.1] | -1.1 [-1.21 to -0.9] | -3.4 [-3.74 to -3.0]

4. Secondary Outcome: Change in Serum Free Testosterone Level
Description: Change in serum free testosterone levels
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin
Number analyzed (Participants) | 66 | 66 | 66
pg/ml | -0.4 [-0.44 to -0.36] | -0.2 [-0.22 to -0.18] | -0.6 [-0.65 to -0.55]

5. Secondary Outcome: Change in Lipid Profile
Description: Change in LDL levels was taken as the indicator of change in lipid profile
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin
Number analyzed (Participants) | 66 | 66 | 66
mg/dl | -10.2 [-11.08 to -9.32] | -8.9 [-9.78 to -8.02] | -20.9 [-22.9 to -18.9]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Cavitation US | Metformin | Cavitation US + Metformin
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 9/66 | 15/66 | 19/66
OTHER ADVERSE EVENTS (reported when occurring in more than 1.52% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cavitation US (N=66) | Metformin (N=66) | Cavitation US + Metformin (N=66)
Gastrointestinal upset (Gastrointestinal disorders) | 0 (0) | 11 (34) | 9 (31)
Generalized malaise (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (19) | 3 (17)
Localized reaction (Skin and subcutaneous tissue disorders) | 9 (19) | 0 (0) | 7 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes